CLINICAL TRIAL: NCT00997152
Title: A Phase II, Randomized, Double-Blind, Placebo-controlled, Multi-Center, Parallel Group Study Evaluating the Efficacy, Safety and Pharmacokinetics of JTT-654 Administered for 12 Weeks in Untreated or Metformin-treated Type 2 Diabetic Patients
Brief Title: Efficacy and Safety Study of JTT-654 in Type 2 Diabetic Patients
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Akros Pharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AT654-U-09-004
Record Dates: First submitted 2009-10-14; First posted 2009-10-19 (Estimated); Last update posted 2013-02-04 (Estimated); Status verified 2013-01

CONDITIONS: Type II Diabetes Mellitus
Keywords: Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Dose 1 JTT-654 (Experimental)
  Interventions: Drug: JTT-654
- Dose 2 JTT-654 (Experimental)
  Interventions: Drug: JTT-654
- Placebo (Placebo Comparator)
  Interventions: Drug: JTT-654 Placebo

INTERVENTIONS:
Drug: JTT-654 — Tablets
  Arms: Dose 1 JTT-654; Dose 2 JTT-654
Drug: JTT-654 Placebo — Tablets
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the effect of JTT-654 on diabetes as well as the safety, tolerability and pharmacokinetics of JTT-654 in type 2 diabetic patients.

ELIGIBILITY:
Inclusion Criteria:

1. Have type 2 diabetes;
2. Body mass index (BMI) of ≤ 45.0 kg/m2;
3. Are either untreated with respect to hypoglycemic agents OR are currently being treated with a stable dose of metformin alone.

Exclusion Criteria:

1. Females who are pregnant or breast-feeding;
2. Known medical history or presence of type 1 diabetes or pancreatitis, acute metabolic diabetic complications, presence of unstable or rapidly progressing retinopathy, nephropathy or neuropathy;
3. Acute coronary syndrome or uncontrolled hypertension;
4. Does not meet all diet or previous/concomitant medication restrictions criteria, as described in the protocol.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2009-09; Primary Completion 2010-03 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Change in Fasting Plasma Glucose (FPG) levels | 3 months

SECONDARY OUTCOMES:
Change in glycosylated hemoglobin (HbA1c) levels | 3 months
Effect on glycated albumin, insulin, C-peptide, glucagon and lipid parameters | 3 months
Safety (biochemistry, hematology, urinalysis and adrenal-related markers) and tolerability (adverse events) | 3 months

CONTACTS AND LOCATIONS:
Locations (42):
- United States (42):
  - Birmingham, Alabama
  - Chandler, Arizona
  - Phoenix, Arizona
  - Tempe, Arizona
  - Chino, California
  - Greenbrae, California
  - Huntington Park, California
  - Los Angeles, California
  - Paramount, California
  - Sacramento, California
  - Walnut Creek, California
  - West Covina, California
  - DeLand, Florida
  - Hialeah, Florida
  - Hollywood, Florida
  - Jacksonville, Florida
  - Miami, Florida
  - Port Orange, Florida
  - Marietta, Georgia
  - Addison, Illinois
  - Chicago, Illinois
  - Indianapolis, Indiana
  - Oxon Hill, Maryland
  - New Bedford, Massachusetts
  - Great Falls, Montana
  - Charlotte, North Carolina
  - Morehead City, North Carolina
  - Cincinnati, Ohio
  - Marion, Ohio
  - Oklahoma City, Oklahoma
  - Lansdale, Pennsylvania
  - Bristol, Tennessee
  - Carrollton, Texas
  - Corpus Christi, Texas
  - Dallas, Texas
  - Houston, Texas
  - Katy, Texas
  - San Antonio, Texas
  - Sugar Land, Texas
  - Norfolk, Virginia
  - Richmond, Virginia
  - Virginia Beach, Virginia